CLINICAL TRIAL: NCT02674178
Title: FSH/LH Ratio as a Predictor of IVF Outcome in Young and Older Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Maged, Assistant professor, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 145
Record Dates: First submitted 2016-01-31; First posted 2016-02-04 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Invitro Fertilization

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Age <35 (Active Comparator): < 35 years old included 201 women who are further subdivided according o FSH/LH ratio into G1A (201 patients) with FSH/LH ratio <2 and G1B (37 patients) with FSH/LH ratio ≥2.
  Interventions: Procedure: Invitro fertilization
- Age ≥ 35 (Active Comparator): . Group 2 ≥ 35 years old included 34 women who are further subdivided according o FSH/LH ratio into G2A (25 patients) with FSH/LH ratio <2 and G2B (9 patients) with FSH/LH ratio ≥2
  Interventions: Procedure: Invitro fertilization

INTERVENTIONS:
Procedure: Invitro fertilization — All participants underwent long protocol. Daily SC injection of Triptorelin 0.1 mg started at day 21 of the cycle prior to stimulation cycle and continued till the day of hCG injection. Gn stimulation started in a starting dose of 150-300 IU/day depending on patients age and previous gonadotropin response. then the dose was adjusted according to ovarian response monitored by serum E2 and ultrasound evaluation. All patients were followed up by Transvaginal ultrasound scan daily or on alternate days
  Triggering by HCG 10000 IU IM when at least 2 follicles reached a mean diameter of 18 mm [18]
  Ovum pick-up (OPU) was done 34-36 hours after hCG injection Transfer of cleaving embryos was done on day 3 after oocyte retrieval

SUMMARY:
All women had normal uterine cavity determined by previous hysterosalpingography or hysteroscopy. Women with abnormally low Gn as hypothalamic hypogonadism , High LH as PCOS and women with abnormal endocrine functions as abnormal thyroid or adrenal functions were excluded. Any woman with ovarian cyst or azopermic male partner was also excluded.

The patients were subjected to history taking, including age, duration, type and cause of infertility and medical history. Full examination including general and abdominal and vaginal examination was done followed by ultrasound evaluation for presence of 3 or more pre-antral follicles and exclusion of ovarian cysts.

Basal day 3 hormonal evaluation for FSH, LH and E2 in a natural cycle was done. E2, FSH and LH levels were determined using Immulite system (Siemens Healthcare diagnostics,UK).The intra- and inter-assay coefficients of variation were 15% and 16% for E2, 4.8% and 26% for LH. FSH analytical sensitivity was 0.1 mIU/ml.

All participants underwent long protocol. Daily SC injection of Triptorelin : Decapeptyl 0.1 mg (Ferring, Switzerland) 0.1 mg started at day 21 of the cycle prior to stimulation cycle and continued till the day of hCG injection. Gn stimulation started after fulfilling stimulation start criteria of thin endometrium < 5 mm and low E2 < 50 and LH < 5IU/l [18] with either HMG(Menogon; Ferring, Switzerland) or rFSH (Gonal-f; Merck Serono, Germany) in a starting dose of 150-300 IU/day depending on patients age and previous gonadotropin response. then the dose was adjusted according to ovarian response monitored by serum E2 and ultrasound evaluation. All patients were followed up by Transvaginal ultrasound scan daily or on alternate days according to the ovarian response to treatment starting on treatment cycle day (6) for folliculometry and endometrial thickness and pattern.

Triggering by HCG 10000 IU IM (Pregnyl, Organon, the Netherlands) when at least 2 follicles reached a mean diameter of 18 mm [18]

Cycle cancellation was decided when transvaginal ultrasound scan on cycle day (9) revealed no adequate follicular growth (<3 mature follicles).

Ovum pick-up (OPU) was done 34-36 hours after hCG injection under transvaginal ultrasound guide.

DETAILED DESCRIPTION:
All women had normal uterine cavity determined by previous hysterosalpingography or hysteroscopy. Women with abnormally low Gn as hypothalamic hypogonadism , High LH as PCOS and women with abnormal endocrine functions as abnormal thyroid or adrenal functions were excluded. Any woman with ovarian cyst or azopermic male partner was also excluded.

The patients were subjected to history taking, including age, duration, type and cause of infertility and medical history. Full examination including general and abdominal and vaginal examination was done followed by ultrasound evaluation for presence of 3 or more pre-antral follicles and exclusion of ovarian cysts.

Basal day 3 hormonal evaluation for FSH, LH and E2 in a natural cycle was done. E2, FSH and LH levels were determined using Immulite system (Siemens Healthcare diagnostics,UK).The intra- and inter-assay coefficients of variation were 15% and 16% for E2, 4.8% and 26% for LH. FSH analytical sensitivity was 0.1 mIU/ml.

All participants underwent long protocol. Daily SC injection of Triptorelin : Decapeptyl 0.1 mg (Ferring, Switzerland) 0.1 mg started at day 21 of the cycle prior to stimulation cycle and continued till the day of hCG injection. Gn stimulation started after fulfilling stimulation start criteria of thin endometrium < 5 mm and low E2 < 50 and LH < 5IU/l [18] with either HMG(Menogon; Ferring, Switzerland) or rFSH (Gonal-f; Merck Serono, Germany) in a starting dose of 150-300 IU/day depending on patients age and previous gonadotropin response. then the dose was adjusted according to ovarian response monitored by serum E2 and ultrasound evaluation. All patients were followed up by Transvaginal ultrasound scan daily or on alternate days according to the ovarian response to treatment starting on treatment cycle day (6) for folliculometry and endometrial thickness and pattern.

Triggering by HCG 10000 IU IM (Pregnyl, Organon, the Netherlands) when at least 2 follicles reached a mean diameter of 18 mm [18]

Cycle cancellation was decided when transvaginal ultrasound scan on cycle day (9) revealed no adequate follicular growth (<3 mature follicles).

Ovum pick-up (OPU) was done 34-36 hours after hCG injection under transvaginal ultrasound guide.

Metaphase II ocytes were analyzed. ICSI procedure was performed in all cases. Fertilization was assessed 16-18 h after ICSI and embryo quality was evaluated 2 and 3 days after ICSI was determined according to the number of blastomeres and the degree of fragmentation and multinucleation[19]. Oocytes were collected and embryos were cultured in ISM1culture medium (Origio medicult media, Denmark).

Transfer of cleaving embryos was done on day 3 after oocyte retrieval (using Labotect semi-rigid catheter; labotect GmbH, Germany) All patients received luteal support in the form of daily progesterone (Prontogest, Amsa, Italy) 100 mg IM daily starting from day of ovum retrieval [18] till day of hCG testing. Serum β hCG level was assessed on day 14 after ET .

The primary outcome parameters evaluated were clinical pregnancy (defined as the presence of gestational sac containing fetal hearts on ultrasound scan). Other parameters included occurrence of multiple pregnancy, Abortion and ectopic cases per pregnancies, dose of Gn, duration of stimulation, E2 and Progesterone levels at day of HCG triggering, endometrial thickness at day of HCG triggering, number of follicles > 16 mm , number of retrieved follicles , number of oocytes fertilized, number of good ET and cancellation rate.

The participants were divided according to age into 2 groups: Group 1<35 years old who are further subdivided according to FSH/LH ratio into G1A with FSH/LH ratio <2 and G1B with FSH/LH ratio ≥2. Group 2 ≥ 35 years old who are further subdivided according o FSH/LH ratio into G2A with FSH/LH ratio <2 and G2B with FSH/LH ratio ≥2. The use of cutoff value is supported by previous studies [20,21]

ELIGIBILITY:
Inclusion Criteria:

* less than 41 years old , with normal menstrual cycle with a range of 24 - 35 days with day 3 FSH less than 10 mIU/ml in natural cycle and normal serum prolactin . All women had normal uterine cavity determined by previous hysterosalpingography or hysteroscopy

Exclusion Criteria:

* Women with abnormally low Gn as hypothalamic hypogonadism , High LH as PCOS and women with abnormal endocrine functions as abnormal thyroid or adrenal functions were excluded. Any woman with ovarian cyst or azopermic male partner was also excluded.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 235 (Actual)
Dates: Start 2012-06; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
clinical pregnancy | 14 days after embryo transfer
  the presence of gestational sac containing fetal hearts on ultrasound scan

SECONDARY OUTCOMES:
multiple pregnancy | 14 days after embryo transfer
Abortion cases per pregnancies | 12 weeks after ET
ectopic cases per pregnancies | 4 weeks after ET

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, MD, Principal Investigator — Kasr Alainy medical school
Locations (1):
- Kasr Alainy medical school, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No